CLINICAL TRIAL: NCT04689269
Title: Endobronchial Intubation With the King Vision and McGrath Laryngoscopes in Simulated Easy and Difficult Airways by Novices. (eKingMath)
Brief Title: Learning Curve of Endobronchial Intubation Using Video Laryngoscopes
Acronym: eKingMath
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB-PGS-2020-01-390
Record Dates: First submitted 2020-12-25; First posted 2020-12-30 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Endobronchial Intubation

STUDY DESIGN:
Intervention Model Description: A single-center, interventional, crossover, single-blind (participant), prospective, trial in simulated "easy" and "difficult" airway. The study will be conducted according to Good Clinical Practice (GCP) Guidelines and abide by the principles of the Declaration of Helsinki.
Who Masked: Participant
Masking Description: Participants will be blind to the data collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- McGrath-King Vision (Active Comparator): The participants will attempt double-lumen tube intubation using the McGrath (X-blade) laryngoscope then they will use the King Vision (channelled blade size 3) in the same order.
  Interventions: Other: The simulated "easy" airway; Other: The simulated "difficult" airway; Device: King Vision Laryngoscope; Device: MacGrath Laryngoscope
- King Vision-McGrath (Active Comparator): The participants will attempt double-lumen tube intubation using the King Vision (channelled blade size 3) then they will use the McGrath (X-blade) laryngoscope in the same order.
  Interventions: Other: The simulated "easy" airway; Other: The simulated "difficult" airway; Device: King Vision Laryngoscope; Device: MacGrath Laryngoscope

INTERVENTIONS:
Other: The simulated "easy" airway — A high-fidelity simulator (Airway Management Trainer, model AA-3100, Laerdal Medical Ltd., Orpington, England, UK) will be equipped to create an easy airway situation by adjusting the manikin until it becomes in a neutral position
Other: The simulated "difficult" airway — A high-fidelity simulator (Airway Management Trainer, model AA-3100, Laerdal Medical Ltd., Orpington, England, UK) will be equipped to create a "difficult" airway scenario will be established by placing the occiput on an Oasis Elite™ Prone Head Rest, Adult (140 mm in height) (Covidien, Mansfield, MA, USA), and inhibiting head and neck movement by securing the head with an adhesive tape, simulating the effect produced by a cervical-collar.
Device: King Vision Laryngoscope — Using a King Vision Laryngoscope for placement of the DLT
Device: MacGrath Laryngoscope — Using a MacGrath Laryngoscope for placement of the DLT

SUMMARY:
The use of video laryngoscopes for endobronchial intubation has its own potential benefits particularly in case of airway difficulty. It is not clear how many cases are required to show competency in successful endobronchial intubation using McGrath and King Vision video laryngoscopes in simulated "easy" and "difficult" airways by novices.

The here proposed randomized crossover clinical trial will test the learning curve of using each of McGrath and King Vision video laryngoscopes in simulated "easy" and "difficult" airways with respect to the number of intubation trials for successful endobronchial intubation

DETAILED DESCRIPTION:
Surgeries that require lung isolation have been using double-lumen tubes (DLT) for endobronchial intubation as the preferred method due to its numerous advantages.

However, the larger diameter of the DLT compared to the single-lumen tube can be more difficult to insert during intubation. [1] The use of video laryngoscopes (VL), which were found to have lower rates of intubation failure, reduced incidences of tracheal and laryngeal trauma, improved glottic view, and increased ease of use, are gaining interest for its use in endobronchial intubation. [2, 3]

The use of McGrath® VL systems for DLT endobronchial intubation has been studied and compared to that of conventional laryngoscopy, as well as that of other VL systems. When compared to the conventional Macintosh laryngoscope, McGrath® VL has been consistently associated with a better glottic visualization. [4 - 6] Other advantages include reduced need for external laryngeal manipulation and a lower rate of intubation-associated complications, such as bronchospasm and trauma to the oral mucosa. [7] However, results regarding time to intubation have been controversial.

The use of King Vision® VL for DLT endobronchial intubation has not been studied as much as the McGrath® video laryngoscope. Two studies compared the King Vision® VL system to the conventional Macintosh laryngoscope and to other VL systems. When comparing King Vision® to Macintosh laryngoscope, the time to intubation was comparable between the two devices. [8, 9] However, one study found that in a simulated easy airway, a significantly longer time to intubation was shown with King Vision® VL. [9] King Vision® VL and Macintosh laryngoscope were also comparable in terms of glottic visualization, intubation difficulty, first-pass success rates, need for optimizing maneuvers, and postoperative symptoms indicative of pharyngeal or laryngeal trauma. [8, 9]

Therefore, competency in endobronchial intubation using video aided laryngoscopes is built through continuous and regular hands-on training. [10] The learning curve of the novice is usually monitored aiming to detect when satisfactory performances are reached. This is widely done using the cumulative sum analysis (CUSUM) test, which provides an objective evaluating method of skill learning via ongoing monitoring. [11]

* Educational Course.

  * All participants will attend a 30-minutes didactic virtual training course on the Zoom platform equipped with a slide presentation including a demonstrative video on the endobronchial intubation and the tips and tricks for using the two study devices.
  * Additionally, a 5-minute hands-on practice session would be provided on each simulated airway model under close supervision by the investigators (AK, MK, SS, and TAG).
* Before each DLT intubation attempt, the manikin, laryngoscope blade, and DLT will be lubricated.
* After completing the DLT intubation, participants should have a 15-minute break before performing intubation using another laryngoscope.
* All intubations will be performed with a 35-Fr left-side DLT.
* The participants will not be allowed to watch each other to avoid any learning effect through observation.

DATA ANALYSIS

Updated and finalized statistical analysis plan will be written, before closing the database.

ELIGIBILITY:
Inclusion Criteria:

* Novice medical school students in using the devices tested.
* Are not familiar with double-lumen tube (DLT) insertion.
* Having no previous experience with the two tested video laryngoscopes for tracheal intubation.

Exclusion Criteria:

* Decline consent to participate.
* No written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
The learning curve of using the device tested | through study completion, an average of 1 month
  The learning curve will be measured with the successful endobronchial intubation within 180 seconds on simulated "easy" and "difficult" airways using McGrath and King Vision video laryngoscopes by cumulative sum (CUSUM) analysis using an EXCEL Spreadsheet.
  Performance of the participants will be assessed for the duration of the study until completing 25 intubation attempts on each of the simulated "easy" and "difficult" airway models with a minimum of one day apart from each model. 25 intubation attempts

SECONDARY OUTCOMES:
Time to endobronchial intubation | for 180 seconds from the passage of the video laryngoscope through the central incisors
  The time needed to achieve endobronchial intubation, which starts from the passage of the video laryngoscope through the central incisors to when the tip of the bronchial lumen passes through the glottis, as confirmed by the investigator through the display screens.
Time to placement of the endobronchial tube | for 360 seconds from the passage of the video laryngoscope through the central incisors
  The time to placement of the endobronchial tube in the left main bronchus
Percentage of glottic opening (POGO) score | for 180 seconds from the passage of the video laryngoscope through the central incisors
  The best view during laryngoscopy using the classification described by percentage of glottic opening (POGO) score
The difficulty of intubation | for 180 seconds from the passage of the video laryngoscope through the central incisors
  The difficulty of intubation evaluated using a visual analog scale (VAS) (ranging from 0, meaning extremely easy, to 100, which is extremely difficult).
The first-pass success | for 360 seconds from the passage of the video laryngoscope through the central incisors
  The first-pass success ratio is calculated as the number of first-attempt successes over the number of intubation attempts.
The number of times the video laryngoscope is withdrawn from mouth | for 180 seconds from the passage of the video laryngoscope through the central incisors
  The number of times the video laryngoscope is withdrawn from mouth then inserted again.
The number of times optimization maneuvers | for 180 seconds from the passage of the video laryngoscope through the central incisors
  The number of times optimization maneuvers are used in each attempt
The number of required external laryngeal manipulation | for 180 seconds from the passage of the video laryngoscope through the central incisors
  The number of required external laryngeal manipulation to improve the glottic view
The preferred device | For 4 weeks from the start of study
  The preferred device as rated by the participant after completing all intubation attempts

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Khidr, MD, Principal Investigator — Assistant Professor & Consultant of Anesthesia and Surgical Intensive Care; Mohamed M El Tahan, MD, Study Chair — Professor of Cardiothoracic Anaesthesia & Surgical Intensive Care
Locations (1):
- Imam Abdulrahman Bin Faisal University, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) will be available to other researchers on request for 3 years after completing the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: for 3 years after completing the study.
Access Criteria: Upon an official request sent to the principal investigator.

REFERENCES:
- [Background] Russell T, Slinger P, Roscoe A, McRae K, Van Rensburg A. A randomised controlled trial comparing the GlideScope((R)) and the Macintosh laryngoscope for double-lumen endobronchial intubation. Anaesthesia. 2013 Dec;68(12):1253-8. doi: 10.1111/anae.12322. PMID 24219251
- [Background] Lewis SR, Butler AR, Parker J, Cook TM, Schofield-Robinson OJ, Smith AF. Videolaryngoscopy versus direct laryngoscopy for adult patients requiring tracheal intubation: a Cochrane Systematic Review. Br J Anaesth. 2017 Sep 1;119(3):369-383. doi: 10.1093/bja/aex228. PMID 28969318
- [Background] Risse J, Schubert AK, Wiesmann T, Huelshoff A, Stay D, Zentgraf M, Kirschbaum A, Wulf H, Feldmann C, Meggiolaro KM. Videolaryngoscopy versus direct laryngoscopy for double-lumen endotracheal tube intubation in thoracic surgery - a randomised controlled clinical trial. BMC Anesthesiol. 2020 Jun 16;20(1):150. doi: 10.1186/s12871-020-01067-x. PMID 32546128
- [Background] Yao WL, Wan L, Xu H, Qian W, Wang XR, Tian YK, Zhang CH. A comparison of the McGrath(R) Series 5 videolaryngoscope and Macintosh laryngoscope for double-lumen tracheal tube placement in patients with a good glottic view at direct laryngoscopy. Anaesthesia. 2015 Jul;70(7):810-7. doi: 10.1111/anae.13040. Epub 2015 Feb 27. PMID 25721326
- [Background] Yoo JY, Park SY, Kim JY, Kim M, Haam SJ, Kim DH. Comparison of the McGrath videolaryngoscope and the Macintosh laryngoscope for double lumen endobronchial tube intubation in patients with manual in-line stabilization: A randomized controlled trial. Medicine (Baltimore). 2018 Mar;97(10):e0081. doi: 10.1097/MD.0000000000010081. PMID 29517671
- [Background] Bakshi SG, Gawri A, Divatia JV. McGrath MAC video laryngoscope versus direct laryngoscopy for the placement of double-lumen tubes: A randomised control trial. Indian J Anaesth. 2019 Jun;63(6):456-461. doi: 10.4103/ija.IJA_48_19. PMID 31263297
- [Background] El-Tahan MR, Khidr AM, Gaarour IS, Alshadwi SA, Alghamdi TM, Al'ghamdi A. A Comparison of 3 Videolaryngoscopes for Double-Lumen Tube Intubation in Humans by Users With Mixed Experience: A Randomized Controlled Study. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):277-286. doi: 10.1053/j.jvca.2017.08.009. Epub 2017 Aug 4. PMID 29056498
- [Background] El-Tahan MR, Al'ghamdi AA, Khidr AM, Gaarour IS. Comparison of three videolaryngoscopes for double-lumen tubes intubation in simulated easy and difficult airways: a randomized trial. Minerva Anestesiol. 2016 Oct;82(10):1050-1058. Epub 2016 May 12. PMID 27171733
- [Background] Failor E, Bowdle A, Jelacic S, Togashi K. High-fidelity simulation of lung isolation with double-lumen endotracheal tubes and bronchial blockers in anesthesiology resident training. J Cardiothorac Vasc Anesth. 2014 Aug;28(4):865-9. doi: 10.1053/j.jvca.2013.07.015. Epub 2013 Nov 12. PMID 24231196
- [Background] Altun D, Ozkan-Seyhan T, Camci E, Sivrikoz N, Orhan-Sungur M. Learning Curves for Two Fiberscopes in Simulated Difficult Airway Scenario With Cumulative Sum Method. Simul Healthc. 2019 Jun;14(3):163-168. doi: 10.1097/SIH.0000000000000368. PMID 30908421